CLINICAL TRIAL: NCT03618797
Title: A Multicenter, Randomized, Double-blinded, Parallel, Therapeutic Confirmatory Clinical Trial to Evaluate the Efficacy and Safety of Pitavastatin Versus Pitavastatin/Fenofibrate in Complex-dyslipidemia Patients
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Pitavastatin/Fenofibrate in Complex-dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL-PIF-301
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Complex-dyslipidemia
MeSH Terms: interventions — Fenofibrate; pitavastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HL-PIF cap.160/2mg + Placebo (Experimental): * Fenofibrate pellet (as micronized fenofibrate 160mg) and Pitavastatin Ca 2mg
  * once a day
  Interventions: Drug: HL-PIF cap.160/2mg + Placebo
- Livalo tab. 2mg + Placebo (Active Comparator): * Pitavastatin ca 2mg
  * once a day
  Interventions: Drug: Livalo tab. 2mg + Placebo

INTERVENTIONS:
Drug: HL-PIF cap.160/2mg + Placebo — Fenofibrate pellet (as micronized fenofibrate 160mg) and Pitavastatin Ca 2mg
  Other Names: Fenofibrate 160mg/Pitavastatin Ca 2mg
  Arms: HL-PIF cap.160/2mg + Placebo
Drug: Livalo tab. 2mg + Placebo — Pitavastatin ca 2mg
  Other Names: Pitavastatin Ca 2mg
  Arms: Livalo tab. 2mg + Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Pitavastatin versus Pitavastatin/Fenofibrate in complex-dyslipidemia patients.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the efficacy of the Pitavastatin/Fenofibrate in complex-dyslipidemia patients by the reduction of non-HDL-Cholesterol levels compared with Pitavastatin.

ELIGIBILITY:
Inclusion Criteria:

* High risk patient to Coronary Heart Disease
* At visit 1(Screening)

  1. If treated with Pitavastatin 2mg monotherapy 4 weeks prior to this study : LDL-C<100mg/dL and 150mg/dL≤TG<500mg/dL, randomize without run-in period
  2. If non treated with Pitavastatin 2mg monotherapy 4 weeks prior to this study : LDL-C≥100mg/dL and 150mg/dL≤TG<500mg/dL, treatment of Pitavastatin 2mg for 4 weeks(run-in period)
* LDL-C<100mg/dL and 150mg/dL≤TG<500mg/dL after 4 weeks of Pitavastatin 2mg monotherapy

Exclusion Criteria:

* Subject with acute artery disease
* Subject with congestive heart failure(NYHA class III~IV) or uncontrolled arrhythmia
* Secondary or iatrogenic dyslipidemia caused by hypothyroidism, nephrotic syndrome etc.
* AST or ALT > 2XULN, Serum Creatinine > 2.5mg/dL, Creatinine phosphokinase > 2XULN
* Subject with gall bladder disease or pancreatitis
* Uncontrolled hypertension
* Endocrine or metabolic disease affected on serum lipid or liprotein
* Subject with medical history of myopathy or rhabdomyolysis caused by Statin treatment, hereditary myopathy or family history
* Not eligible to participate for the study at the discretion of investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The mean percentage change of Non-HDL Cholesterol | from baseline at week 8
  Change rate of Non-HDL-C after 8 weeks compared to baseline (%)

SECONDARY OUTCOMES:
The mean percentage change of Non-HDL Cholesterol | from baseline at week 4
  Change rate of Non-HDL-C after 4 weeks compared to baseline (%)
The mean percentage change of LDL-C | from baseline at week 4,8
  Change rate of LDL-C after 4 and 8 weeks compared to baseline (%)
The mean percentage change of HDL-C | from baseline at week 4,8
  Change rate of HDL-C after 4 and 8 weeks compared to baseline (%)
The mean percentage change of LDL-C/HDL-C | from baseline at week 4,8
  Change rate of LDL-C/HDL-C after 4 and 8 weeks compared to baseline (%)
The mean percentage change of TC/HDL-C | from baseline at week 4,8
  Change rate of TC/HDL-C after 4 and 8 weeks compared to baseline (%)
The mean percentage change of non-HDL-C/HDL-C | from baseline at week 4,8
  Change rate of non-HDL-C/HDL-C after 4 and 8 weeks compared to baseline (%)
The mean percentage change of VLDL-C | from baseline at week 4,8
  Change rate of VLDL-C after 4 and 8 weeks compared to baseline (%)
The mean percentage change of TG | from baseline at week 4,8
  Change rate of TG after 4 and 8 weeks compared to baseline (%)
The mean percentage change of TC | from baseline at week 4,8
  Change rate of TC after 4 and 8 weeks compared to baseline (%)
The mean percentage change of Apo Al | from baseline at week 4,8
  Change rate of Apo Al after 4 and 8 weeks compared to baseline (%)
The mean percentage change of Apo B | from baseline at week 4,8
  Change rate of Apo B change after 4 and 8 weeks compared to baseline (%)
The mean percentage change of Apo Al/Apo B | from baseline at week 4,8
  Change rate of Apo Al/Apo B after 4 and 8 weeks compared to baseline (%)
The mean percentage change of fibrinogen | from baseline at week 4,8
  Change rate of fibrinogen after 4 and 8 weeks compared to baseline (%)
The mean percentage change of hs-CRP | from baseline at week 4,8
  Change rate of hs-CRP after 4 and 8 weeks compared to baseline (%)
Achievement rate(%) of treatment goals after 4 weeks and 8 weeks | from baseline at week 4,8
  LDL-C<100mg/dL & non-HDL-C <130mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bae Seung, Principal Investigator — The Catholic University of Korea

REFERENCES:
- [Derived] Ihm SH, Chung WB, Lee JM, Hwang BH, Yoo KD, Her SH, Song WH, Chae IH, Park TH, Kim JH, Jeon DW, Cho BR, Kang SH, Park SD, Lee JB, Woo JT, Lee BW, Han KA, Won KH, Kim HS, Yu JM, Chung CH, Kim HJ, Cho HC, Seung KB. Efficacy and Tolerability of Pitavastatin Versus Pitavastatin/Fenofibrate in High-risk Korean Patients with Mixed Dyslipidemia: A Multicenter, Randomized, Double-blinded, Parallel, Therapeutic Confirmatory Clinical Trial. Clin Ther. 2020 Oct;42(10):2021-2035.e3. doi: 10.1016/j.clinthera.2020.08.002. Epub 2020 Sep 2. PMID 32891418